CLINICAL TRIAL: NCT07084675
Title: Impact of Mild Dehydration and Subsequent Rehydration on Cellular Stress and Physiological Performance
Brief Title: Dehydration, Rehydration, and Impact on Physiology
Acronym: DRIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Principal Investigator, Hui Ying Luk, Assistant Professor, Texas Tech University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB2025-288
Record Dates: First submitted 2025-07-03; First posted 2025-07-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Aging
Keywords: rehydration; hypohydration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydration-Dehydration-Rehydration (HDR) Protocol Arm (Experimental): Participants in this arm complete the HDR Protocol over 12 days and attend five lab visits.
  Interventions: Behavioral: Hydration-Dehydration-Rehydration Protocol (HDR)

INTERVENTIONS:
Behavioral: Hydration-Dehydration-Rehydration Protocol (HDR) — The HDR Protocol is a 12-day, sequential fluid manipulation intervention designed to assess the physiological effects of controlled changes in hydration status. The protocol consists of three consecutive 4-day phases:
  Hydration Phase (Days 1-4): Participants follow a standardized fluid intake protocol designed to promote and maintain a euhydrated state. Hydration status is monitored using objective measures such as urine specific gravity and body mass.
  Dehydration Phase (Days 5-8): Participants adhere to a fluid-restriction regimen to induce a hypohydrated state. The level of dehydration is verified through the same hydration status measures to ensure consistent and safe hypohydration.
  Rehydration Phase (Days 9-12): Participants resume the standardized fluid intake protocol used during the Hydration Phase to restore euhydration. Rehydration effectiveness is confirmed through repeated hydration assessments.

SUMMARY:
Our goal is to determine whether hydration status influences inflammation, and overall physiological performance in adults aged 45-65.

Aim 1: The effects of 4-day mild dehydration followed by 4-day rehydration (defined as approximately 2-3% body mass loss) on H2O2, upstream inflammatory signal (NFkB), mitochondrial fragmentation, and autophagy in circulating PBMCs.

Aim 2: The effects of 4-day mild dehydration followed by 4-day rehydration (defined as approximately 2-3% body mass loss) on fasting glucose, sleep performance, and strength performance.

Participant will:

complete a 4-day hydration protocol, followed by a 4-day dehydration protocol, and then a 4-day rehydration protocol.

attend five laboratory visits for testing: Day 1: Informed consent and familiarization Day 2: Pre-hydration testing (before the 4-day hydration protocol) Day 3: Pre-dehydration testing (before the dehyration protocol) Day 4: Post-dehydration testing (after the dehydration protocol) Day 5: Post-rehydration testing (after the rehydration protocol)

ELIGIBILITY:
Inclusion Criteria:

* Apparently Healthy
* BMI < 30 kg/m2
* Body weight is at least 110 lbs

Exclusion Criteria:

* Currently pregnant
* Have Type 1 Diabetes or Type 2 Diabetes
* Have chronic kidney disease or a history of kidney stones
* Have hypertension
* Take medications that can cause fluid retention, such as corticosteroids, chronic use of Nonsteroidal Anti-inflammatory Drugs (NSAIDs), Hormonal Therapies (e.g., estrogen, androgens or anabolic steroids), Antihypertensives, Psychiatric Medications (e.g., Lithium), Vasodilators
* Take medications that reduce fluid retention: diuretics, and RAAS Inhibitors (e.g., ACE inhibitors and ARBs)

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose (mg/dL) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Fasting blood glucose will be measured via fingerstick at each testing visit. Values will be used to examine changes in glucose regulation in response to hydration status across the HDR Protocol phases.
Total body water (L) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Bioelectrical impedance spectroscopy (BIS) will be used to assess changes in total body water, BIS measurements will be collected at each testing visit to evaluate fluid shifts.
Intracellular water (L) | Time Frame: Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Description: Bioelectrical impedance spectroscopy (BIS) will be used to assess changes in intracellular water across hydration phases. BIS measurements will be collected at each testing visit to evaluate fluid shifts.
Extracellular water (L) | Time Frame: Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Description: Bioelectrical impedance spectroscopy (BIS) will be used to assess changes in extracellular water across hydration phases. BIS measurements will be collected at each testing visit to evaluate fluid shifts.
Hand grip strength (kg) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Handgrip strength will be measured using a handheld dynamometer at four time points during the HDR Protocol. Measurements will be used to assess the impact of hydration status on upper body muscular strength.
Isometric leg pull strength (kg) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Isometric lower body strength will be evaluated using a standardized leg pull test at four timepoints during the HDR Protocol. Results will be used to determine the effect of hydration status on lower body muscular strength.
Total sleep time (hrs) | through study completion, 18 days
  Total sleep time will be continuously monitored throughout the HDR Protocol using a wearable device.
Sleep efficiency (%) | through study completion, 18 days
  Sleep efficiency will be continuously monitored throughout the HDR Protocol using a wearable device.
Number of awakenings (count) | through study completion, 18 days
  Number of awakenings will be continuously monitored throughout the HDR Protocol using a wearable device.
PBMC H2O2 ( µg/mL) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Peripheral blood mononuclear cells (PBMCs) will be isolated from whole blood samples collected at four time points during the HDR Protocol. H2O2 will be assessed.
DRP1 (Arbitrary Units) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Peripheral blood mononuclear cells (PBMCs) will be isolated from whole blood samples collected at four time points during the HDR Protocol. Fission expression (DRP1).
MFN (Arbitrary Units) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Peripheral blood mononuclear cells (PBMCs) will be isolated from whole blood samples collected at four time points during the HDR Protocol. Mitochondrial fusion expression (MFN) will be assessed.
PINK1 (Arbitrary Units) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Peripheral blood mononuclear cells (PBMCs) will be isolated from whole blood samples collected at four time points during the HDR Protocol. Mitophagy marker (PINK1) will be assessed.
Parkin (Arbitrary Units) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Peripheral blood mononuclear cells (PBMCs) will be isolated from whole blood samples collected at four time points during the HDR Protocol. Mitophagy marker (Parkin) will be assessed.
Malondialdehyde (nmol/mg) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Peripheral blood mononuclear cells (PBMCs) will be isolated from whole blood samples collected at four time points during the HDR Protocol. Lipid peroxidation will be assessed by measuring malondialdehyde concentrations.

SECONDARY OUTCOMES:
Change in hydration status via urine specific gravity (USG) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Hydration status will be assessed using urine specific gravity (USG) at four time points across the HDR Protocol: prior to the hydration phase, following the hydration phase, after the dehydration phase, and after the rehydration phase. These values will be used to confirm the effectiveness of each fluid manipulation phase.
Total lean mass (g) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Body composition will be assessed using dual-energy X-ray absorptiometry (DXA) at four time points across the HDR Protocol. Total lean mass will be evaluated in relation to hydration status at each phase.
Total fat mass (g) | Day 2 (Pre-hydration testing), Day 3 (Pre-dehydration testing), Day 4 (Post-dehydration testing), Day 5 (Post-rehydration testing)
  Body composition will be assessed using dual-energy X-ray absorptiometry (DXA) at four time points across the HDR Protocol. Total fat mass will be evaluated in relation to hydration status during each phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All raw data generated from this project will be stored on cloud-based servers at Texas Tech University. Cleaned data in an analysis-ready format will be stored in REDCap and periodically uploaded to repositories. Data of sufficient quality from human participants will be uploaded the Aging Research Biobank to allow others to validate replicate research findings.
  In alignment with the Data Submission Worksheet for the Aging Research Biobank, the following will be submitted to accompany deidentified data derived from human participants:
  * Full study protocol
  * Names and descriptions of data sets
  * Manual of operations
  * Annotated data collection forms
  * Data dictionary
  * Documentation of calculated variables
  * Summary of deidentification and crosslinking of study ID with new randomized ID
  * Any changes made to the protocol over time
  * Frozen datasets used for the primary publication, when applicable